CLINICAL TRIAL: NCT06296875
Title: Uncovering the Mechanisms Through Which Krill Oil Increases Muscle Function in Older Adults.
Brief Title: The Krill Ageing Muscle Mechanisms (KAMM) Study
Acronym: KAMM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Stuart Gray, Professor of Muscle and Metabolic Health, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KAMM
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Sarcopenia
Keywords: Krill oil; Muscle Strength; Neuromuscular function; Physical function
MeSH Terms: conditions — Sarcopenia | interventions — Plant Oils

STUDY DESIGN:
Intervention Model Description: 1:1 parallel group design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All supplements will be matched for taste and look
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vegetable oil (Placebo Comparator): 4g/day vegetable oil for 24 weeks
  Interventions: Dietary Supplement: Vegetable oil
- Krill oil (Active Comparator): 4/g/day krill oil for 24 weeks
  Interventions: Dietary Supplement: Krill oil

INTERVENTIONS:
Dietary Supplement: Vegetable oil — mixed vegetable oil
  Arms: Vegetable oil
Dietary Supplement: Krill oil — Krill oil
  Other Names: (SuperbaBoost)
  Arms: Krill oil

SUMMARY:
This study aims to determine the mechanisms via which krill oil supplementation increases muscle strength and whether this translates to improvements in gait and functional characteristics in older adults. The studies we will carry out will establish, in healthy older adults, the effects of 6 months of supplementation with krill oil

Objective 1) Muscle structure and function Hypothesis: Krill oil supplementation will increase muscle size and strength alongside positive changes in muscle architecture (pennation angle and fascicle length).

Objective 2) Neuromuscular control and central nervous system (CNS) function Hypothesis: Krill oil supplementation will improve Neuromuscular Junction (NMJ) transmission stability and increase central drive and intramuscular coherence, as a measure of muscle synergy.

Objective 3) Gait and functional characteristics Hypothesis: Krill oil supplementation will improve gait and functional characteristics.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) </= 30 kg/m2
* Age >/= 65 years
* Capacity to consent
* Living within the Glasgow area

Exclusion Criteria:

* Diabetes mellitus
* Severe cardiovascular disease
* Seizure disorders
* Uncontrolled hypertension (>150/90mmHg)
* Active cancer or cancer that has been in remission <5 years
* Participation in any resistance exercise training within the last 6 months
* Impairments which may limit ability to perform assessments of muscle function
* Dementia
* Fish/shellfish allergy
* Taking medication known to affect muscle (e.g. steroids, Selective serotonin reuptake inhibitors) or anticoagulants (e.g. warfarin)
* Taking omega-3 supplements in the last 3 months
* Regularly consuming 1 or more portions of oily fish per week
* Not able to understand English

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Grip strength | Change from baseline to 24 weeks
  We will measure grip strength using a handgrip dynamometer, making 3 maximal contractions in each hand, with the dominant hand recorded. The highest grip strength will be used in analysis.
Neuromuscular junction transmission instability | Change from baseline to 24 weeks
  We will assess peripheral motor unit (MU) characteristics in the vastus lateralis muscle using intramuscular electromyography
Gait speed | Change from baseline to 24 weeks
  We will measure gait speed using a gaitrite connected mat during a 4 m walk test and the timed up and go test at usual speed.

SECONDARY OUTCOMES:
Knee extensor maximal torque | Change from baseline to 24 weeks
  We will measure the muscle strength of the knee extensor muscles during a maximal voluntary contraction (MVC)
Vastus lateralis muscle cross sectional area | Change from baseline to 24 weeks
  We will measure this using ultrasound
Vastus lateralis pennation angle | Change from baseline to 24 weeks
  We will measure this using ultrasound
Vastus lateralis fascicle length | Change from baseline to 24 weeks
  We will measure this using ultrasound
Erythrocyte fatty acid composition | Change from baseline to 24 weeks
  Blood samples (15 ml each visit) will be collected
Knee extensor force steadiness | Change from baseline to 24 weeks
  During the contractions to measure NMJ transmission instability we will also calculate force steadiness, as a measure of neuromuscular control
Vastus lateralis motor unit conduction velocity | Change from baseline to 24 weeks
  will be measured using High Density surface electromyography (HDsEMG) during submaximal (10%, 30%, 50% and 70% of MVC) and during the MVC
Vastus lateralis and vastus medialis intramuscular coherence | Change from baseline to 24 weeks
  Motor unit spike train will be measured using the surface electromyography (sEMG) electrodes while participants exert 20% of maximum voluntary contraction
Hand flexor muscles intermuscular coherence | Change from baseline to 24 weeks
  Intermuscular coherence will be measured for 1 min on 20% of MVC using sEMG electrodes.
Cortico-muscular coherence between sensory motor cortex and hand extensor muscles | Change from baseline to 24 weeks
  Cortico-muscular coherence is a derived measure, based on measurement of the electroencephalography (EEG) and motor unit spikes. EEG electrodes will be placed over the motor area of hands and worn during hand contractions
Femoral Nerve Stimulation | Change from baseline to 24 weeks
  Single stimuli will be delivered to the muscle while participants maintain a 20% MVC isometric contraction, and the intensity of stimulation was increased until a plateau in twitch amplitude and rectus femoris M-wave (Mmax) occurs. Supramaximal stimulation will then be delivered by increasing the final stimulator output intensity by a further 30%.
Transcranial Magnetic Stimulation (TMS) | Change from baseline to 24 weeks
  Motor evoked potentials (MEPs) will be elicited in the rectus femoris of the dominant leg via single pulse TMS and assessed using electromyographic (EMG) recordings.
TMS Inhibition | Change from baseline to 24 weeks
  corticomotor inhibition during the MVCs a single TMS stimulation will be delivered over the motor cortex.
TMS Excitation | Change from baseline to 24 weeks
  For assessment of corticospinal excitability, participants will maintain a 20% MVC isometric contraction while 20 single TMS pulses, separated by 6 s, will be delivered over the motor cortex
Gait characteristics during 4m walk test and the timed up and go test | Change from baseline to 24 weeks
  The 4 m walk test involves participants walking a 4m distance at a normal walking pace, walking through the 4m line at the end of the gaitrite mat. The Timed Up and Go test (timed version of the Get Up and Go test) involves the participant sitting on a chair getting up, walking 3 meters in front of them across the gaitrite mat, returning to the chair and sitting down. The Theia markerless system will be used to extract Gait parameters
Gait cycle with leg support parameters | Change from baseline to 24 weeks
  We will also get posture information from the 3D skeleton measurements and balance (pitch and roll) which are important in assessing fall risks and functional gait.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No